CLINICAL TRIAL: NCT03441737
Title: The Effects of Acute Aerobic Exercise on Inhibitory Control in Temporarily Abstinent Smokers
Brief Title: Aerobic Exercise and Inhibitory Control
Acronym: AMIAEIC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not receive funding to support this project.
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Dr. Harry Prapavessis, Principal Investigator, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1795AM
Record Dates: First submitted 2018-02-09; First posted 2018-02-22 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Smoking Cessation; Inhibition (Psychology)
Keywords: Aerobic exercise; Antisaccades; Urge to Smoke; Adults
MeSH Terms: conditions — Smoking Cessation; Inhibition, Psychological | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Aerobic exercise intervention
  Interventions: Behavioral: Exercise
- Non-Exercise (Active Comparator): Non-aerobic exercise intervention
  Interventions: Behavioral: Non-Exercise

INTERVENTIONS:
Behavioral: Exercise — 20 minutes of aerobic exercise (walking on a treadmill) at 2/3 of participant's maximum heart rate (maximum heart rate calculated as 220-age).
  Arms: Exercise
Behavioral: Non-Exercise — 20 minutes of sitting in the laboratory with access to magazines and the internet.
  Arms: Non-Exercise

SUMMARY:
Although more than half of Canadian smokers in 2015 attempted to quit, with one-third attempting more than once, successful smoking cessation (quitting) remains a challenge. Relapse (return to smoking) has been attributed to failures in inhibitory control. Inhibitory control is the ability to suppress actions. Previous studies have identified that aerobic exercise improves inhibitory control and reduces the urge to smoke. This study will examine whether an acute bout of moderate intensity aerobic exercise (i.e. brisk walk on a treadmill) will improve inhibitory control, increase time to first cigarette smoked, and reduce urges to smoke during a brief period of abstinence. Inhibitory control will be assessed using the antisaccade task, which requires the participant to shift their gaze away from a visual target presented to them. Phase I will include assessments of smoking behaviours, physical activity levels, urges to smoke, and inhibitory control. Phase II will consist of a 12-hour smoking abstinence period conducted at home, followed by reassessment of urges to smoke and inhibitory control. Participants will then be randomized to either 20 minutes of aerobic exercise or sitting. Following the intervention, reassessment of urges to smoke, inhibitory control, and time to first cigarette smoked will be conducted.

DETAILED DESCRIPTION:
The participant will be provided a letter of information and an informed consent form. Once they have signed the informed consent form, the following procedures will take place:

Phase I:

* Initial biological confirmation of carbon monoxide reading: Participant will briefly blow air into a Smokelyzer (device which assesses how much carbon monoxide in parts per million is present in the breath of a smoker)
* Baseline questionnaires: Participant will be asked to fill out to the best of their ability the following questionnaires:

  1. Demographic questionnaire (Asks you identifiable information concerning, your age, email telephone number)
  2. Smoking history questionnaire ("What is the approximate date and time of the last cigarette you have smoked?")
  3. Fagerstrom Test for Nicotine Dependence ("How many cigarettes do you smoke each day?")
  4. Godin Leisure-Time Exercise Questionnaire ("In the last 7 days, how many times have you completed mild intensity exercise for 15 minutes or more?")
  5. Physical Activity Readiness Questionnaire ("Do you feel pain in your chest at rest?")
  6. Urge to Smoke ("I have an urge for a cigarette")
  7. Heart rate will be measured with a heart rate monitor. Blood pressure will be measured with an electronic blood pressure cuff.
* Cognitive computer task: Participant will be asked to complete a computer task which assesses inhibitory control (the cognitive ability to suppress responses to stimuli). The Antisaccade Task will be used to assess inhibitory control in this study.

Phase II:

* Smoking abstinence period: The participant will be instructed at the end of Phase I that they will have to complete a 12 hour smoking abstinence period (refraining from smoking cigarettes or consumption of any tobacco products) at home before coming back into the lab. The participant will be also notified that the co-investigator will be able to assess whether they completed this abstinence period through assessing the carbon monoxide reading on the Smokelyzer.
* Biological confirmation of carbon monoxide reading: Participant will briefly blow air into a Smokelyzer (device which assess how much carbon monoxide in parts per million is present in the breath of a smoker). The participant will have to blow below 10 parts per million carbon monoxide to have successfully abstained and thus participate in Phase II.
* Questionnaire: Participant will be asked to fill out to the best of their ability the following questionnaire:

  f. Urge to Smoke ("I have an urge for a cigarette")
* Cognitive Computer Task: Participant will complete the same Antisaccade Task as outlined in Phase I.
* Intervention Participant will be randomly assigned (through a randomly generated number sequence) to either 20 minutes of aerobic exercise or 20 minutes of sitting.
* Aerobic Exercise Intervention: The participant will complete a 20 minute walking exercise on a treadmill.
* Non Exercise: The participant will be in a seated position in the lab waiting room. They will be provided with magazines and computer access.
* Post Intervention:
* Questionnaire: Participant will be asked to fill out to the best of their ability the following questionnaire:

  f. Urge to Smoke ("I have an urge for a cigarette")

The participant will then be told to notify the co-investigator of when they light their next cigarette through a time-stamped email or text message. The time in minutes from when they leave the lab (time: 0) until the message is received will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years of age
* Smoke at least 10 cigarettes per day (or more) for at least 6 months
* Able to perform a twenty-minute exercise task at a moderate intensity (2/3 of participant's maximum heart rate) without health implications
* Can read and write in English
* Have email or phone number for contacting purposes

Exclusion Criteria:

* Do not have Chronic Obstructive Pulmonary Disease
* Do not have a medical condition that prevents you from exercise (e.g. heart attack in the past year, heart disease, irregular heartbeat, etc.)
* Do not have history of eye injury or neurological impairment
* Do not have an orthopaedic limitation
* Are not pregnant

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Inhibitory Control | 24 hours post participant start date
  Cognitive computer task: Participant will be asked to complete a computer task which assesses inhibitory control (the cognitive ability to suppress responses to stimuli). The Antisaccade Task will be used to assess inhibitory control in this study. A saccade is a rapid eye movement towards a visual target. An antisaccade is a rapid eye movement away from a visual target. The ability to suppress making an eye movement towards a visual target gauges inhibitory control. The participant will be seated in a chair facing a computer screen in which visual stimuli (a cross) will appear. The participant will be fitted into a chin rest and a monocle will be adjusted so that images of eye movements can be assessed. A training phase will take place at the beginning of the task to familiarize the participant with the instructions. The participant will make a series of saccades and antisaccades. The reaction times and directional errors to the visual stimuli will be recorded.

SECONDARY OUTCOMES:
Urge to Smoke | 24 hours post participant start date
  Questionnaire: 1 item from the Questionnaire of Smoking Urges (QSU) will be used to assess the urge to smoke.
Time to First Cigarette | 24 hours post participant start date
  The time to first cigarette post intervention will be calculated from time 0 being when the participant leaves the lab until the co-investigator receives a time-stamped message from the participant that they have light their first cigarette.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Harry Prapavessis, Principal Investigator — Western University

IPD SHARING:
Plan to Share IPD: No